CLINICAL TRIAL: NCT01282385
Title: Hemodynamic Effect of the Combination of Simvastatin With Non-cardioselective Beta Blockers in Patients With Cirrhosis and Clinically Significant Portal Hypertension
Brief Title: Hemodynamic Effect of Simvastatin With Beta Blockers in Clinical Portal Hypertension
Acronym: SIMBETA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Candido Villanueva, Hospital de la Santa Creu i Sant Pau
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IIBSP-SIM-2010-04
Record Dates: First submitted 2011-01-21; First posted 2011-01-25 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2011-01

CONDITIONS: Liver Cirrhosis; Portal Hypertension.
MeSH Terms: conditions — Liver Cirrhosis; Hypertension, Portal | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- simvasatin (Experimental): a) patients responding to treatment with beta-blockers, in which she was treated with nadolol Subsequently randomized into two treatment arms, double-blind:
  a.1: simvastatin 20 mg capsules, starting at doses of 20 mg / 24 hours, may increase to 40 mg according to clinical and laboratory tolerance.
  a.2: placebo capsules with external characteristics similar to simvastatin.
  b) non-responders to treatment with beta blockers, receive treatment with carvedilol.Subsequently randomized into two treatment arms, double-blind
  b.1: simvastatin 20 mg capsules, starting at doses of 20 mg / 24 hours, may increase to 40 mg according to clinical and laboratory tolerance.
  b.2: placebo capsules with external characteristics similar to simvastatin.
  Interventions: Drug: Simvastatin
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Simvastatin — simvastatin 20 mg capsules, starting at doses of 20 mg / 24 hours, may increase to 40 mg according to clinical and laboratory tolerance
  Arms: simvasatin
Drug: placebo — placebo capsules with external characteristics similar to simvastatin administrated each 24 hours.
  Arms: placebo

SUMMARY:
In the genesis and maintenance of PH associated with liver cirrhosis are two mechanisms that act synergistically. The first is an increase in hepatic vascular resistance, due in part to the disruption of liver structure inherent cirrhosis, and increased hepatic vascular tone is caused by the contraction of perivascular smooth muscle cells, myofibroblasts and hepatic stellate cells, which represents about 30% of global intrahepatic resistance and is believed to be due to the production Defective nitric oxide (NO). The second mechanism, which maintains and exacerbates HTP, is an increase of splanchnic blood flow caused by increased NO and other vasodilators at this level

In this regard, we believe that in patients with compensated liver cirrhosis, with portal pressure gradient> 10 mmHg, both acute responders betablockers test as non-responders, the association of antifibrotic drugs and / or vasodilators, chronic liver selective May be beneficial in the control of portal hypertension

DETAILED DESCRIPTION:
This study was prospective, randomized, controlled, double blind, in which patients who met the inclusion criteria and give written consent to participate in the study underwent a baseline hemodynamic study to determine the portal pressure gradient (GPSH). During the event, will assess the acute response to intravenous administration of propranolol. It is considered good hemodynamic response to declining GPSH >20% from baseline or decrease to <12 mmHg. At the conclusion of the baseline hemodynamic study patients will be divided into 2 treatment groups:

a) patients responding to treatment with beta-blockers, in which she was treated with nadolol at doses of 40mg/24horas (increasing the dose every 2-3 days as tolerated, to a maximum of 240 mg / 24 hours. Subsequently randomized into two treatment arms, double-blind:

a.1: simvastatin 20 mg capsules, starting at doses of 20 mg / 24 hours, may increase to 40 mg according to clinical and laboratory tolerance.

a.2: placebo capsules with external characteristics similar to simvastatin.

b) non-responders to treatment with beta blockers, carvedilol receive treatment with an initial dose of 6.25 mg / 24 hours, may increase to 25mg/dia if good clinical tolerance (HR and BP monitoring) and analytical (renal function and electrolyte disturbances) . Subsequently randomized into two treatment arms, double-blind b.1: simvastatin 20 mg capsules, starting at doses of 20 mg / 24 hours, may increase to 40 mg according to clinical and laboratory tolerance.

b.2: placebo capsules with external characteristics similar to simvastatin.

In order to evaluate the long-term hemodynamic effect, patients will receive treatment for a month and hemodynamic study will be repeated to completion.

ELIGIBILITY:
Inclusion Criteria:

* Liver cirrhosis diagnosed by previous biopsy or by clinical, laboratory, ultrasound,
* PPG> 10 mmHg,
* Presence of large esophageal varices or small varices with red spots, varices of any size and Pugh C, and / or gastric fundic varices of any size, in a recent gastroscopy (<1 month)
* Absence of previous episodes of gastrointestinal bleeding
* Written informed consent.

Exclusion Criteria:

* Age <18 and> 80 years;
* Episode of variceal bleeding,
* Thrombosis splenoportal axis,
* Hepatocarcinoma,
* Terminal liver failure (Child-Pugh scale> 13 points);
* Any comorbidity involving a medical drugs and / or a life expectancy <12 months,
* Severe chronic renal insufficiency (creatinine> 150 g / L),
* Absolute contraindication or allergy treatment with statins to simvastatin;
* Concomitant potent inhibitors of CYP3A4 (eg., itraconazole, ketoconazole, inhibitors of HIV protease, erythromycin, clarithromycin, telithromycin and nefazodone),
* Pretreatment (<1 month) or other lipid-lowering with simvastatin,
* Previous episodes rhabdomyolysis;
* Contraindication to beta-blockers (COPD with bronchial hyperresponsiveness, aortic stenosis, AV block, intermittent claudication, severe psychosis, bronchial asthma),
* Hypersensitivity to beta blockers,
* Concomitant administration of potent inhibitors of cytochrome P-450 (quinidine, fluoxetine, paroxetine, and propafenone)
* Active alcoholic hepatitis,
* Refusal to participate in the study or the informed consent claim;
* Pre-treatment with beta blockers or nitrates, or endoscopic treatment for varicose veins or portosystemic shunts;
* Pregnancy and lactation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-04; Primary Completion 2014-04 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
improvement of the hemodynamic response rate | 1 month.
  The main objective is to assess whether, in patients with compensated cirrhosis, portal pressure greater than 10mmHg and esophageal varices at risk, the association of a liver selective vasodilator and simvastatin together with non-cardioselective beta blockers can improve the hemodynamic response rate.

SECONDARY OUTCOMES:
Portal hypertension complications. | 1 month
  Development of complications related to portal hypertension (gastrointestinal bleeding related to portal hypertension, ascites, hepatic encephalopathy).
Adverse effects | 1 month
  adverse effects related to medication

CONTACTS AND LOCATIONS:
Overall Officials: Candido Villanueva, MD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona, Spain

REFERENCES:
- [Background] Bosch J. Carvedilol for portal hypertension in patients with cirrhosis. Hepatology. 2010 Jun;51(6):2214-8. doi: 10.1002/hep.23689. No abstract available. PMID 20513005
- [Background] Trebicka J, Hennenberg M, Laleman W, Shelest N, Biecker E, Schepke M, Nevens F, Sauerbruch T, Heller J. Atorvastatin lowers portal pressure in cirrhotic rats by inhibition of RhoA/Rho-kinase and activation of endothelial nitric oxide synthase. Hepatology. 2007 Jul;46(1):242-53. doi: 10.1002/hep.21673. PMID 17596891
- [Result] Abraldes JG, Albillos A, Banares R, Turnes J, Gonzalez R, Garcia-Pagan JC, Bosch J. Simvastatin lowers portal pressure in patients with cirrhosis and portal hypertension: a randomized controlled trial. Gastroenterology. 2009 May;136(5):1651-8. doi: 10.1053/j.gastro.2009.01.043. Epub 2009 Jan 24. PMID 19208350
- [Result] Tripathi D, Therapondos G, Lui HF, Stanley AJ, Hayes PC. Haemodynamic effects of acute and chronic administration of low-dose carvedilol, a vasodilating beta-blocker, in patients with cirrhosis and portal hypertension. Aliment Pharmacol Ther. 2002 Mar;16(3):373-80. doi: 10.1046/j.1365-2036.2002.01190.x. PMID 11876689